CLINICAL TRIAL: NCT03909659
Title: A Randomized-Controlled Trial to Determine the Effects on Blood Pressure of A Reduced-sodium Added-potassium Salt Substitute Among Adults With Hypertension in India
Brief Title: The Effects on Blood Pressure of Salt Substitute Among Adults With Hypertension in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SSiIS
Record Dates: First submitted 2019-03-31; First posted 2019-04-10 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Normal salt
- Reduced-sodium added-potassium salt substitute (Experimental): salt substitute
  Interventions: Behavioral: Dietary sodium reduction

INTERVENTIONS:
Behavioral: Dietary sodium reduction — A supply of a reduced-sodium added-potassium salt substitute
  Arms: Reduced-sodium added-potassium salt substitute

SUMMARY:
Blood pressure is a key modifiable risk factor for cardiovascular disease in India. Drug therapies are highly effective and are recommended by local guidelines to reduce the risks of serious cardiovascular complications. Behavioural approaches to blood pressure control based upon sodium reduction are also recommended but there are no interventions proven effective in India.

Mean sodium intake in India is about 5g/day (equivalent to about 12.5g salt) which is, more than double World Health Organization (WHO) recommendations. Reduced sodium, added potassium salt substitutes have favourable effects on blood pressure in settings where discretionary salt use is high, but have not been tested in India. This single-site, Salt Substitute on blood pressure in India Study will investigate the effects of reduced sodium added potassium salt substitution on blood pressure in rural areas where hypertension is a prevalent disease problem and additional, scalable and affordable interventions are required. The primary objective is to assess the effects of salt substitute on SBP at 3 months follow-up. The secondary objectives are to determine effects on DBP, urinary sodium and potassium levels and to determine acceptability of the salt substitute.

The study will be a double-blinded, randomized-controlled trial done in the Hyderabad region amongst adult volunteers with a history of hypertension diagnosed by a health professional. The main exclusion criteria will be known serous kidney disease or use of potassium containing medications by the individual or others living in the household. Written informed consent will be obtained from potential participants followed by baseline data collection. Eligible individuals will then be assigned at random to receive double-blind salt or salt substitute which will be used to replace all dietary salt used for cooking and seasoning over the next 3 months. Follow-up will be at one and three months after randomisation for blood pressure, urinary electrolytes and acceptability of the intervention.

DETAILED DESCRIPTION:
Excess sodium intake is associated with high blood pressure which is a leading risk for cardiovascular disease (CVD) in India. Drug therapies are highly effective interventions for blood pressure lowering and are recommended by local guidelines to reduce the risks of serious cardiovascular complications. Behavioural approaches to blood pressure control based upon sodium reduction are also recommended but there are no interventions proven effective and sustainable in India.

Mean sodium intake in India is about 5g/day (equivalent to about 12.5g salt) which is more than double World Health Organization (WHO) recommendations. Reduced sodium, added potassium salt substitutes have favourable effects on blood pressure in settings where discretionary salt use is high, but have not been tested in India. Salt substitution is of particular interest because it has great potential for scaling in under-served and resource poor settings.

This study will investigate the effects of salt substitution on blood pressure in rural areas where hypertension is a highly prevalent disease problem and additional, scalable and affordable blood pressure lowering interventions are required. Accordingly, the primary objective is to assess the effects of a reduced sodium, added potassium salt substitute compared to usual salt on systolic blood pressure (SBP) at 3-months follow-up. The secondary objectives are to determine effects on diastolic blood pressure (DBP), urinary sodium and potassium levels and to determine acceptability of the salt substitute among patients with hypertension.

The study will be a double-blinded, randomized-controlled trial done in the villages of the Hyderabad district amongst adult volunteers with a self-reported history of hypertension. The main exclusion criteria will be known serous kidney disease or use of potassium containing medications by the individual or others living in the household. Written informed consent will be obtained from potential participants followed by baseline data collection. Eligible individuals will then be assigned at random to receive double-blind salt or salt substitute which will be used to replace all dietary salt required for cooking and seasoning in the household over the next 3-months. Follow-up will be at one and three months after randomisation for assessment of blood pressure and acceptability of the intervention, with urinary electrolytes measured at baseline and 3-months.

The sample size will be 440 participants randomized in a 1:1 ratio to intervention or control which will provide more than 80% power (P=0.05) to detect a 5 mmHg or greater difference in SBP between randomized groups. This estimate assumes a mean of 140mmHg and a standard deviation of 20mmHg for SBP at baseline. We will seek to recruit comparable numbers of men and women. Analyses will be done using the principle of intention-to-treat and a repeated measures analysis of variance that incorporates baseline, 1-month and 3-month measures of SBP to maximize the efficiency of the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or over
* History of hypertension diagnosed by a health professional - hypertension may be self-reported and antihypertensive drugs may or may not be used for management. There is no entry criterion based upon blood pressure measurements made at the baseline survey
* Eat most of their meals in the home
* Consent to participate

Exclusion Criteria:

* Participant or family member is using a potassium-sparing diuretic
* Participant or family member is using a potassium supplement
* Participant or family member has known significant renal dysfunction
* Participant or family member has other reason for concern about use of salt substitute
* Participant is not expected to live longer than 6 months from the date of assessment
* Another member of the household is already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | three months
  As measured by using an automated blood pressure monitor according to established standardized methods.

SECONDARY OUTCOMES:
Diastolic Blood Pressure | three months
  As measured by using an automated blood pressure monitor according to established standardized methods.
Urinary sodium excretion | three months
  A field-based measurement of sodium made using the meter (HORIBA Ltd, Japan), which uses a direct ion-selective electrode technique to measure sodium concentrations.
Urinary potassium excretion | three months
  A field-based measurement of potassium made using the meter (HORIBA Ltd, Japan), which uses a direct ion-selective electrode technique to measure potassium concentrations.
Acceptability of the study salt substitute | three months
  Acceptability of the study salt substitute will be measured using the following questions at baseline and follow-up: How many days in the last week did you use study salt? If you were meant to use the study salt in the last week but did not use it every day, what is the reason? If you use the study salt in the last week: How did you use it? How many meals did you use the study salt during the day? Did you enjoy the taste? (1 = disliked a lot; 10 = liked a lot)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yu, Principal Investigator — The George Institute; Thout Sudhir Raj, Principal Investigator — The George Institute
Locations (1):
- The George Institute for Glaobal Health India, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu J, Thout SR, Li Q, Tian M, Marklund M, Arnott C, Huffman MD, Praveen D, Johnson C, Huang L, Pettigrew S, Neal B, Wu JHY. Effects of a reduced-sodium added-potassium salt substitute on blood pressure in rural Indian hypertensive patients: a randomized, double-blind, controlled trial. Am J Clin Nutr. 2021 Jul 1;114(1):185-193. doi: 10.1093/ajcn/nqab054. PMID 33782684